CLINICAL TRIAL: NCT05668546
Title: Is Isokinetic Knee Muscle Strength an Indicator of Total Knee Arthroplasty
Brief Title: Is Isokinetic Testing an Indicator of Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Ilknur Saral, Ass. Prof., Bahçeşehir University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: 395
Record Dates: First submitted 2022-12-08; First posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Knee Osteoarthritis
Keywords: arthroplasty; diagnostic x-ray; knee; muscle strength dynamometer; visual analog scale
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: After the surgical decision was made, the patients were referred to the physiatrist by the orthopedist without informing which knee would be operated on. The physiatrist and the patient did not know which knee would be operated, so the tests were performed blindly.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgical knee group (Experimental): This study analyzed 58 knees of 29 unilateral TKA candidates, divided into the surgical and non-surgical knee groups
  Interventions: Device: isokinetic testing CSMI HUMAC NORM instrument
- non surgical knee group (Experimental): This study analyzed 58 knees of 29 unilateral TKA candidates, divided into the surgical and non-surgical knee groups
  Interventions: Device: isokinetic testing CSMI HUMAC NORM instrument

INTERVENTIONS:
Device: isokinetic testing CSMI HUMAC NORM instrument — The strength (PT) of the bilateral knee flexors and extensors were tested with isokinetic test. Tests were performed under the guidance of a rehabilitation medicine specialist, and the system was calibrated prior to their commencement. The patients were seated in upright position and were fixed with pelvic and thigh belts. Concentric extension (PT_E) and concentric flexion (PT_F) were measured between the 0° and 90° knee ranges at angular velocities of 60°/s and 180°/s (60 PT_E, 60 PT_F, 180 PT_E, and 180 PT_F, respectively) The tests were repeated five times at each velocity, and the highest PTs were selected for statistical analysis. The participants performed repeated trials before sets, while a 20-second rest was provided between sets.

SUMMARY:
In this study, investigators analyzed whether the isokinetic knee muscle strength of patients undergoing unilateral total knee arthroplasty (TKA) is a predictor for surgery.

Patients and Methods: In total, 29 unilateral TKA candidates (58 knees; mean age = 66.69 ± 7.42 years; mean symptom duration = 10 ± 5.40 years) were enrolled. The knees of patients with bilateral advanced knee osteoarthritis (stage 3 or 4), according to the Kellgren-Lawrence (K-L scale), that were scheduled for unilateral TKA were divided into surgical and non-surgical groups. An isokinetic testing system was used to assess knee flexor and extensor muscle strength (peak torque) at angular velocities of 60°/s and 180°/s (five cycles per velocity). The radiological (X-ray-based K-L scale and magnetic resonance imaging (MRI)-based quadriceps angle) and clinical findings (isokinetic test and visual analog scale pain scores) in both groups were compared. The isokinetic test results correlated with the radiological findings of the surgery group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced (Kellgren-Lawrence stage 3 or 4) bilateral knee osteoarthritis (OA).
* Unilateral total knee replacement surgery recommended by orthopedics according to pain status

Exclusion Criteria:

* Neurological diseases that could affect knee muscle strength
* Rheumatological diseases
* Diagnosis of osteoarthritis below 3 according to Kellgren-Lawrence classification

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Knee flexion and extension muscle strengths assessed by isokinetic dynamometer | cross-sectional study, baseline
  In the isokinetic evaluation, both 60 PT_E (Peak Torque _Extension) and 60 PT_F (Peak Torque_Flexion) were evaluated.The tests were repeated five times at each velocity, and the highest PTs were selected for statistical analysis. The participants performed repeated trials before sets, while a 20-second rest was provided between sets.
Osteoartritis gradings assessed by Kellgren-Lawrence grading system | cross sectional study, baseline
  Kellgren-Lawrence grading system was used. Each radiograph was assigned a grade from 0 to 4, which correlated to increasing severity of OA, with Grade 0 signifying no presence of OA and Grade 4 signifying severe OA
Pain assessed by Visual analog scale | cross sectional study, baseline
  The visual analog scale (VAS) pain score of each individual was also recordedThe Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). Investigators asked the patient to rate their current level of pain by placing a mark on the line.
Quadriceps angle | cross sectional study, baseline
  Q angle of knees were recorded. It is defined as the angle formed between the quadriceps muscles and the patella tendon.The Q angle measured in standing. Normal Q angle score for females is between 13-18° and in males is between 12-15°, with values greater than and lesser these are considered abnormal

CONTACTS AND LOCATIONS:
Overall Officials: ilknur saral, Ass Prof, Principal Investigator — Bahcesehir University, Department of Health Sciences
Locations (1):
- Memorial Sisli Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 3 months after publication